CLINICAL TRIAL: NCT03935373
Title: Using the DNA Exome Sequencing Tools to Explore the Association Among Gene Sequence, TCM Pattern, TCM Tongue Diagnosis and TCM Pulse Diagnosis for Sjögren's Syndrome
Brief Title: DNA Exome Sequencing TCM for Sjögren's Syndrome
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017-09-006C#3
Record Dates: First submitted 2019-04-22; First posted 2019-05-02 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Sjögren's Syndrome
Keywords: Immune regulation; Sjögren's syndrome; Gene modulation; Traditional Chinese Medicine pattern; Traditional Chinese Medicine tongue diagnosis; Traditional Chinese Medicine pulse diagnosis; Proteomics; Oral microbiome
MeSH Terms: conditions — Sjogren's Syndrome | interventions — Microbiota; Base Sequence; Th1-Th2 Balance; Liver Function Tests; Kidney Function Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 1. The DNA of Sjögren's syndrome patients and health subjects will take to do the DNA Exome sequencing.
  2. The saliva of Sjögren's syndrome patients and health subjects will take to do the oral microbiome.
  3. The protein of Sjögren's syndrome patients and health subjects will take to do the proteomics.
  4. The RNA of Sjögren's syndrome patients and health subjects will store to do the RNA sequencing.
  5. The plasma of Sjögren's syndrome patients and health subjects will store to do the cytokine detection in the future.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sjögren's syndrome: Sjögren's syndrome patients were screened in the rheumatology outpatient departments and Center for Traditional Medicine at Taipei Veterans General Hospital, and were enrolled with the inclusion criteria: (1) primary or secondary SS; (2) aged between 20 and 75 years; (3) fulfilled the 2002 American-European Consensus Criteria for SS (AECG); (4) had no abnormal findings of immune, liver, kidney, or blood function evaluations. And the exclusion criteria were: (1) a history of alcohol abuse, diabetes mellitus, or major life-threatening condition; (2) pregnancy or breastfeeding; or (3) steroid pulse therapy within three months prior to the commencement of our study.
  Interventions: Diagnostic Test: DNA Exome sequencing; Diagnostic Test: Oral microbiome; Diagnostic Test: Proteomics; Diagnostic Test: RNA sequencing; Diagnostic Test: Cytokine; Diagnostic Test: Traditional Chinese Medicine pattern; Diagnostic Test: Traditional Chinese Medicine tongue diagnosis; Diagnostic Test: Traditional Chinese Medicine pulse diagnosis; Diagnostic Test: Heart rate variability; Diagnostic Test: Schirmer's test; Diagnostic Test: Blood function test, liver function test, kidney function test, and immune function test
- Health subjects: Health subjects were screened in the rheumatology outpatient departments and Center for Traditional Medicine at Taipei Veterans General Hospital, and were enrolled with the inclusion criteria: (1) aged between 41 and 63 years (which the age could match the SS patients enrolling in the SS-1 trial); (2) had no chronic inflammatory illness. And the exclusion criteria were: (1) a history of alcohol abuse, diabetes mellitus, or major life-threatening condition; (2) pregnancy or breastfeeding; (3) abnormal findings of immune, liver, kidney, or blood function evaluations; (4) total sleeping time insufficiency less than 6 hours before one day of enrollment; (5) ever took the conventional medicine or hormone within one month; (6) ever encountered the acute illness, allergy reaction, immune, or rheumatic disease within one month.
  Interventions: Diagnostic Test: DNA Exome sequencing; Diagnostic Test: Oral microbiome; Diagnostic Test: Proteomics; Diagnostic Test: RNA sequencing; Diagnostic Test: Cytokine; Diagnostic Test: Traditional Chinese Medicine pattern; Diagnostic Test: Traditional Chinese Medicine tongue diagnosis; Diagnostic Test: Traditional Chinese Medicine pulse diagnosis; Diagnostic Test: Heart rate variability; Diagnostic Test: Blood function test, liver function test, kidney function test, and immune function test

INTERVENTIONS:
Diagnostic Test: DNA Exome sequencing — The DNA of Sjögren's syndrome patients and health subjects will take to do the DNA Exome sequencing.
Diagnostic Test: Oral microbiome — The saliva of Sjögren's syndrome patients and health subjects will take to do the oral microbiome.
Diagnostic Test: Proteomics — The protein of Sjögren's syndrome patients and health subjects will take to do the proteomics.
Diagnostic Test: RNA sequencing — The RNA of Sjögren's syndrome patients and health subjects will store to do the RNA sequencing.
Diagnostic Test: Cytokine — The serum of Sjögren's syndrome patients and health subjects will store to do the cytokine detection in the future.
Diagnostic Test: Traditional Chinese Medicine pattern — Sjögren's syndrome patients and health subjects will take the Traditional Chinese Medicine pattern.
Diagnostic Test: Traditional Chinese Medicine tongue diagnosis — Sjögren's syndrome patients and health subjects will take the Traditional Chinese Medicine tongue diagnosis.
Diagnostic Test: Traditional Chinese Medicine pulse diagnosis — Sjögren's syndrome patients and health subjects will take the Traditional Chinese Medicine pulse diagnosis.
Diagnostic Test: Heart rate variability — Sjögren's syndrome patients and health subjects will take the heart rate variability.
Diagnostic Test: Schirmer's test — Sjögren's syndrome patients will take the Schirmer's test.
  Groups: Sjögren's syndrome
Diagnostic Test: Blood function test, liver function test, kidney function test, and immune function test — Sjögren's syndrome patients and health subjects will take the blood function test (WBC, RBC, Hb, HCT, Platelet, MCV, MCH, and MCHC), liver function test (AST and ALT), kidney function test (BUN and Cre), and immune function test (RF, Anti-SSA, Anti-SSB Ab, ESR, and CRP)

SUMMARY:
To explore the association among gene, TCM pattern, TCM tongue diagnosis and TCM pulse diagnosis with the DNA Exome sequencing tools for Sjögren's syndrome

DETAILED DESCRIPTION:
Objective: To explore the association among gene, TCM pattern, TCM tongue diagnosis and TCM pulse diagnosis with the DNA Exome sequencing tools for Sjögren's syndrome

Method:

This study wants to establish the reference value of DNA gene variants of healthy control for comparing with the Sjögren's syndrome subjects. And the investigators want to use the DNA Exome sequencing tools, proteomics and oral microbiome to explore the association of gene expression between at least 30 Sjögren's syndrome subjects and at least 10 healthy control subjects. Finally, the investigators also analyze the association among gene expression, proteomics and oral microbiome, TCM pattern, TCM tongue diagnosis, TCM pulse diagnosis, and heart rate variability (HRV) for this purpose.

Expected Results:

1. To evaluate the difference among TCM pattern, TCM tongue diagnosis, TCM pulse diagnosis, and HRV for the Sjögren's syndrome and healthy control.
2. To evaluate the immunity-related gene expression for the Sjögren's syndrome and healthy control.
3. To evaluate the proteomics for the Sjögren's syndrome and healthy control.
4. To evaluate the oral microbiome for the Sjögren's syndrome and healthy control.
5. To evaluate the association among the immunity-related gene expression, SSA, SSB and RF.

Keyword: Sjögren's syndrome, Immune regulation, Gene modulation, TCM pattern, TCM tongue diagnosis, TCM pulse diagnosis, proteomics, oral microbiome

ELIGIBILITY:
Sjögren's syndrome

Inclusion Criteria:

* (1) primary or secondary SS
* (2) aged between 20 and 75 years
* (3) fulfilled the 2002 American-European Consensus Criteria for SS (AECG)
* (4) had no abnormal findings of immune, liver, kidney, or blood function evaluations.

Exclusion Criteria:

* (1)a history of alcohol abuse, diabetes mellitus, or major life-threatening condition
* (2) pregnancy or breastfeeding
* (3) steroid pulse therapy within three months prior to the commencement of our study.

Health Subjects

Inclusion Criteria:

* (1) aged 20 and 75 years
* (2) had no chronic inflammatory illness.

Exclusion Criteria:

* (1) a history of alcohol abuse, diabetes mellitus, or major life-threatening condition
* (2) pregnancy or breastfeeding
* (3) abnormal findings of immune, liver, kidney, or blood function evaluations
* (4) total sleeping time insufficiency less than 6 hours before one day of enrollment
* (5) ever took the conventional medicine or hormone within one month
* (6) ever encountered the acute illness, allergy reaction, immune, or rheumatic disease within one month.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sjögren's syndrome patients and Health subjects were screened in the rheumatology outpatient departments and Center for Traditional Medicine at Taipei Veterans General Hospital.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-05-15 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Immunity-related gene expression | One year
  To evaluate the immunity-related gene expression for the Sjögren's syndrome and healthy control.
  DNA exome combine the GATK (Genome Analysis Toolkit) is a tool for detecting the ratio of immunity-related gene expression.
TCM pattern | One year
  To evaluate the difference of TCM pattern between Sjögren's syndrome and healthy control.
  TCM pattern is a tool for detecting the constitution.
TCM tongue diagnosis | One year
  To evaluate the difference of TCM tongue diagnosis between Sjögren's syndrome and healthy control.
  TCM tongue diagnosis is a tool for detecting tongue expression.
TCM pulse diagnosis | One year
  To evaluate the difference of TCM pulse diagnosis between Sjögren's syndrome and healthy control.
  TCM pulse diagnosis is a tool for detecting pulse of radial artery.
Heart rate variability (HRV) | One year
  To evaluate the difference of Heart rate variability (HRV) between Sjögren's syndrome and healthy control.
  HRV is a tool for detecting the ratio between High-frequency (HF) activity and low-frequency (LF) activity.
Immunity-related proteomics expression | One year
  To evaluate the proteomics for the Sjögren's syndrome and healthy control.
  Proteomics is a tool for detecting the ratio of immunity-related proteomics expression.
Immunity-related microbiome expression | One year
  To evaluate the oral microbiome for the Sjögren's syndrome and healthy control.
  Oral microbiome is a tool for detecting the ratio of immunity-related microbiome expression.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Mao Chang, M.D., Ph.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Ching-Mao Chang, Taipei, Taiwan (r.o.c.), Taiwan

IPD SHARING:
Plan to Share IPD: No